CLINICAL TRIAL: NCT03429231
Title: Observational Study With Food Product to Evaluate the Quality of Life of Healthy Postmenopausal Women Who Take Coenzyme Q-Ubiquinol, Compared With Another Group of the Same Age That Does Not Take coenzymeQ-Ubiquinol
Brief Title: Observational Study to Evaluate the Quality of Life of Healthy Postmenopausal Women Who Take Coenzyme Q-Ubiquinol
Status: Completed | Type: Observational
Sponsor: Dr. Santiago Palacios (Other)
Responsible Party: Sponsor-Investigator, Dr. Santiago Palacios, Principal Investigator, Instituto Palacios
Organization: Instituto Palacios (Other)
Other Study IDs: QUbiquinol17
Record Dates: First submitted 2018-01-16; First posted 2018-02-12 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Group: Women who are taking coenzyme Q and who will continue taking it for 3 months
  Interventions: Dietary Supplement: Coenzima Q - QubiquinolCoenzyme Q - Qubiquinol
- Control Group: Women who are not taking coenzyme Q and who will not take it in the next 3 months

INTERVENTIONS:
Dietary Supplement: Coenzima Q - QubiquinolCoenzyme Q - Qubiquinol — Patients in the active group will take one tablet a day orally
  Groups: Active Group

SUMMARY:
Observational study about quality of life in postmenopausal women taking coenzyme Q compared to another group of women of the same age who do not take it

DETAILED DESCRIPTION:
Observational study to evaluate the subjective assessment performed by healthy postmenopausal women who are taking coenzyme Q for 3 months, compared with other groups of the same characteristics that do not take it

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman between 45 and 65 years old
* Woman who is taking coenzyme Q-Ubiquinol and who will continue taking at least the next 3 months
* Woman not taking Coenzyme Q-Ubiquinol and not going to take it in the next 3 months

Exclusión Criteria:

* Patients with severe mental illness.
* Suspicion or abuse of alcohol or other drugs during the 12 months prior to the selection
* Any other consideration or finding that, in the opinion of the investigator, considers the non-participation of the subject in the study.

Age Groups: Child, Adult, Older Adult
Study Population: Healthy postmenopausal woman between 45 and 65 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quality of Life at 3 months | Baseline and 3 months
  To evaluate the quality of life in healthy postmenopausal women who are taking Coenzyme Q-Ubiquinol for 3 months in comparison with another group that does not take them. The Cervantes Health-Related Quality of Life scale for menopause will be used for this outcome. In that scale next to the 0 and the 5 there are words that describe two opposite answers to the question. Between the 0 and the 5 there are also four boxes numbered 1 to 4. The participants should answer the questions by checking the box that best represents what they think and feel. In other words, they should check 5 if they are completely agree and 0 they are completely disagree. If they are not completely agree or disagree, they should check the boxes in between

SECONDARY OUTCOMES:
Change from Baseline General Health at 3 months | Baseline and 3 months
  Health Scale Euroqol EQ-5D will be used for this outcome
Change from Baseline Mood at three months | Baseline and 3 months
  An analogic scale will be used for this outcome in wich 0 points is the best mood and 10 points is worst mood
Change from Baseline Cramps at three months | Baseline and 3 months
  To assess changes in cramps in patients who had them, a general questionnaire about Cramps will be used to assess mainly the intensity and frequency of crambs. Regarding the intensity 0 is the lower pain and 10 is the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No